CLINICAL TRIAL: NCT06004856
Title: A Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of Orelabrutinib in Adult Patients With Chronic Primary Immune Thrombocytopenia
Brief Title: Evaluate the Efficacy and Safety of Orelabrutinib in Adult Patients With Chronic Primary Immune Thrombocytopenia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICP-CL-00126
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Chronic Primary Immune Thrombocytopenia (ITP)
MeSH Terms: interventions — orelabrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orelabrutinib (Experimental)
  Interventions: Drug: Orelabrutinib
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orelabrutinib — Orelabrutinib once daily (QD)
  Arms: Orelabrutinib
Drug: Placebo — Placebo once daily (QD)
  Arms: Placebo

SUMMARY:
A Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of Orelabrutinib in Adult Patients with Chronic Primary Immune Thrombocytopenia

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have had a detailed understanding of the nature, significance, possible benefits, possible inconveniences, and potential risks of the trial, understood the study procedures, and voluntarily signed a written ICF before the study.
2. Males or females aged from 18 to 80 years (including the marginal values).
3. With a body weight of ≥ 35 kg at screening.
4. In accordance with the diagnosis of chronic (≥ 12 months) ITP
5. Patients who have previously received at least one anti-ITP first-line standard treatment (glucocorticoids and/or intravenous immunoglobulin) cannot maintain efficacy, or relapse, or cannot tolerate standard treatment, or have insufficient response.
6. Females of childbearing potential must use an effective method of contraception during the screening period, throughout the entire trial, and for 90 days after the last administration of the investigational medicinal product (IMP).

Exclusion Criteria:

1. Severe hemorrhage occurred within 4 weeks prior to screening.
2. Subjects suffered from severe ITP at screening and were not eligible for participation in this study as judged by the investigator.
3. Subjects had autoimmune systemic diseases other than ITP unless they would not affect the evaluation of the study results in the judgment of the investigator and sponsor medical monitor.
4. Subjects had multiple immune hemocytopenia.
5. Subjects had inherited thrombocytopenia or secondary ITP.
6. Subjects had a history of arterial or venous thromboembolism within 6 months prior to screening.
7. Received prohibited medications within protocol-specified period before the first dose.
8. Received blood transfusion (including platelet transfusion) within 2 weeks prior to the first dose of the investigational drug.
9. Participated in another study of the investigational drug (and/or investigational device) within 30 days or within 5 half-lives prior to screening (whichever is longer), or is currently participating in another study of the investigational drug (and /or investigational device).
10. The last administration of strong CYP3A inhibitors or strong CYP3A inducers (include food, western medicine, traditional Chinese medicine) is within 14 days (or 5 half-lives, whichever is longer) prior to the first dose, or planned to take a drug or food with a strong inhibition or induction of CYP3A during the study period.
11. Received a major surgery (including splenectomy) or trauma (except biopsy) within 28 days prior to the first dose of the investigational drug, or expected to receive a major surgery during the study treatment period.
12. Received splenectomy and had a prior history of overwhelming post-splenectomy infection (OPSI).
13. Had a history of alcohol or drug abuse currently or within the past 1 year, excepting nicotine and caffeine.
14. Received a COVID-19 vaccine, live vaccine, or live-attenuated vaccine within 1 month prior to screening or during the screening period.
15. Previous exposure to BTK inhibitors.
16. Laboratory results did not meet protocol requirements.
17. Pregnant or lactating women.
18. Subjects whose blood cannot be collected, or who had contraindications for blood collection.
19. Other conditions that were not appropriate for participation in the trial as considered by the investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Durable response rate | Throughout the study period, an average of 6 months

CONTACTS AND LOCATIONS:
Locations (45):
- China (45):
  - The first affiliated hospital of bengbu medical college, Bengbu, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing CHAO-YANG Hospital Capital Medcal University, Beijing, Beijing Municipality
  - Peking university People's Hospital, Beijing, Beijing Municipality
  - Xinqiao Hospital of Army Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Huazhong University of Science and Technology Union Shenzhen Hospital, Shenzhen, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - North China University of Science and Technology Affiliated Hospital, Tangshan, Hebei
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Medical College Of Hust, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Chenzhou First People's Hospital, Chenzhou, Hunan
  - The Central Hospital of Yongzhou, Yongzhou, Hunan
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The first Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital Of Shandong University Dezhou Hospital, Dezhou, Shandong
  - Qilu hospital of shandong university, Jinan, Shandong
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Xi'an Central Hospital, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi’an, Shanxi
  - Shaanxi Provincial People'S Hospital, Xi’an, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Affilated Hospital of Southwest Medical University, Luzhou, Sichuan
  - The Second People's Hospital of Yibin, Yibin, Sichuan
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang Uygur Autonomous Region
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial Hospital of Chinese Medicine, Hangzhou, Zhejiang